CLINICAL TRIAL: NCT05143164
Title: Study of Hydrocolloid Dressing for Peritoneal Dialysis Catheter Exit Site Care in Peritoneal Dialysis Patients - a Pilot Study
Brief Title: Hydrocolloid Dressing for Catheter Exit Site Care in Peritoneal Dialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/2434
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Dialysis Catheter Exit Site Infection
Keywords: peritoneal dialysis; exit-site care; exit-site dressing
MeSH Terms: interventions — Bandages, Hydrocolloid; Gentamicins

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hydrocolloid dressing (Experimental): The intervention group will use the weekly hydrocolloid dressing (Duoderm Extra Thin CGF dressing,10 x 10 cm) for peritoneal dialysis exit-site care
  Interventions: Device: hydrocolloid dressing
- Gentamicin cream (Active Comparator): The control group will apply topical gentamicin cream to catheter exit site daily and cover with normal dressing
  Interventions: Drug: Gentamicin Sulfate, Topical

INTERVENTIONS:
Device: hydrocolloid dressing — Duoderm Extra Thin hydrocolloid dressing will be used to cover the catheter exit-site of participants in the intervention group. The dressing will be changed every 7 days or early if the dressing is no longer adhesive.
  Arms: Hydrocolloid dressing
Drug: Gentamicin Sulfate, Topical — Application of gentamicin to exit site daily
  Arms: Gentamicin cream

SUMMARY:
The study aims to examine the use of hydrocolloid dressing for catheter exit-site care in peritoneal dialysis patients. It is a pilot study, and participants will be randomized to either receiving weekly hydrocolloid dressing or daily topical gentamicin cream for exit-site care in peritoneal dialysis patients.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) related infection is one of the main reasons for patients to discontinue PD therapy. Routine exit-site care is crucial for the prevention of infections, however, daily antibiotics use has been associated with the risk of developing drug-resistant bacteria. Moreover, the burden of daily exit-site care can lead to non-compliance with treatment. Hydrocolloid dressing has been used in the management of acute and chronic wounds and is required to change once weekly, but its use has not been examined in the exit-site wound in PD patients.

The study primarily aims to examine PD-related infection (exit site infection or peritonitis rates) between patients using weekly hydrocolloid dressing (experimental group) and those using daily topical application of gentamicin (control group) for exit-site care in PD patients. Secondary aims include time to the first episode of PD-related infection, technique failure, PD infection-related hospitalization, and adverse events. The study will also assess the acceptability of dressing and quality of life between the two groups.

A total of 60 adult peritoneal dialysis patients will be recruited for the study. Patients will be randomly assigned to either the experimental group or the control group. Participants will be followed up at the 4th, 12th, and 24th week of study. The acceptability of the dressing will be assessed using the treatment acceptability questionnaires. The quality of life will be assessed using the ED 5D-5L questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All adult peritoneal dialysis patients (≥ 21 years old) and are followed up at Singapore General Hospital (SGH)

Exclusion Criteria:

* Patients who are unable to provide valid consent, patients who have known allergy to hydrocolloid dressing, patients who have peritoneal dialysis catheter exit site infection or peritonitis within the past 3 months, patients who have dialysate leak at PD catheter exit site, pregnant women, patients with life-expectancy of < 1 year or patients who are currently involved in another study for peritoneal dialysis catheter exit site care.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peritoneal dialysis (PD)-related infection rate | 24 weeks
  PD-related infection (exit-site /tunnel infection or peritonitis) (episode per patient-year)

SECONDARY OUTCOMES:
Time to the first episode of exit-site/tunnel infection or peritonitis | 24 weeks
  Time to first episode of exit-site/tunnel infection or peritonitis (days)
Peritoneal dialysis infection-related hospitalization rate | 24 weeks
  Hospitalization due to peritoneal dialysis-related infection (episode per patient-year)
Technique failure rate | 24 weeks
  Technique failure is defined as transfer to hemodialysis for >= 30 days (episode per patient-year)
Adverse events | 24 weeks
  Adverse events related to the dressing (local or systemic effects)
Quality of life score using ED 5D 5L questionnaire | at 12th week of study
  Quality of life score using ED 5D 5L questionnaire (numerical scores)
Treatment acceptability | at 12th week of study
  Acceptability of dressing will be measured by treatment acceptability questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No